CLINICAL TRIAL: NCT02062905
Title: A Multi-Center, Randomized, Double-Masked, Vehicle Controlled Phase 2 Study Evaluating the Efficacy and Safety of OTX-DP for the Treatment of Chronic Allergic Conjunctivitis Using a Modified Conjunctival Allergen Challenge Model (CAC™)
Brief Title: OTX-14-001: A Phase 2 Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Chronic Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-14-001
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2017-09

CONDITIONS: Chronic Allergic Conjunctivitis
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- OTX-DP (Experimental): OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use
  Interventions: Drug: Dexamethasone
- PV (Placebo Comparator): PV (placebo drug delivery vehicle)
  Interventions: Other: Placebo Vehicle

INTERVENTIONS:
Drug: Dexamethasone
  Arms: OTX-DP
Other: Placebo Vehicle
  Arms: PV

SUMMARY:
The objective of the study was to evaluate the efficacy and safety of OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use when placed in the canaliculus of the eyelid for the treatment of the signs and symptoms of chronic allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Has a positive history of ocular allergies and a positive skin test reaction to a perennial allergen and a seasonal allergen
* Has a positive bilateral CAC reaction to a perennial allergen within minutes of instillation

Exclusion Criteria:

* History of ocular surgical intervention within the past 3 months
* Presence of an active ocular infection or positive history of an ocular herpetic infection at any visit
* Use any of the following disallowed medications during the period indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- OTX-DP Treatment: OTX-DP (sustained release dexamethasone, 0.4 mg)
  OTX-DP treatment
- Placebo Plug Delivery Vehicle: Placebo Plug with no drug
  Placebo Plug with no drug
Period: Overall Study
Arm/Group | OTX-DP Treatment | Placebo Plug Delivery Vehicle
Started | 35 | 33
Completed | 28 | 31
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-DP Treatment | Placebo Plug Delivery Vehicle | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 30 | 64
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Proprietary Ora Calibra Conjunctival Allergen Challenge Ocular Itching Scale (0 - 4 with 0.5 unit increments allowed; "0" = no itching)
Time Frame: 14 days post insertion
Measure: Mean (Standard Deviation); unit: units on a scale (0 -4)
Arm/Group | OTX-DP Treatment | Placebo Plug Delivery Vehicle
Number analyzed (Participants) | 28 | 31
units on a scale (0 -4)
  3 min (14 days post-insertion) | 1.80 (1.068) | 2.58 (0.823)
  5 min. (14 days post-insertion) | 1.72 (0.998) | 2.70 (0.865)
  7 min. (14 days post-insertion) | 1.65 (0.989) | 2.53 (0.880)

2. Secondary Outcome: Conjunctival Redness
Description: Proprietary Ora Calibra Ocular Hyperemia Scale (0 - 4 with 0.5 unit increments allowed; "0" = no redness)
Time Frame: 14 days post insertion
Measure: Mean (Standard Deviation); unit: units on a scale (0 - 4)
Arm/Group | OTX-DP Treatment | Placebo Plug Delivery Vehicle
Number analyzed (Participants) | 28 | 31
units on a scale (0 - 4)
  7 min. (14 days post-insertion) | 1.60 (0.753) | 2.11 (0.727)
  15 min. (14 days post-insertion) | 1.53 (0.753) | 2.23 (0.708)
  20 min. (14 days post-insertion) | 1.54 (0.739) | 2.21 (0.696)

ADVERSE EVENTS:
Arm/Group | OTX-DP Treatment | Placebo Plug Delivery Vehicle
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/33
Other Adverse Events (participants affected / at risk) | 1/31 | 2/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-DP Treatment (N=31) | Placebo Plug Delivery Vehicle (N=33)
depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-DP Treatment (N=31) | Placebo Plug Delivery Vehicle (N=33)
eye discharge (Eye disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other